CLINICAL TRIAL: NCT02906241
Title: PACCT: Partnering Around Cancer Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Eggly (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Susan Eggly, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-098; R01CA200718-01 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: African Americans; prostate cancer; Minority; Racial /Ethnic disparity; Cancer care; patient-physician communication; cancer clinical trial accrual
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients--Intervention (Experimental): Patients are randomized to an intervention group. They participate in all aspects of the study and also receive the intervention, which consists of a booklet.
  Interventions: Behavioral: Patients: Questions to Ask Your Doctor: A Workbook for Patient-Doctor Teams
- Patients--Usual Care (No Intervention): Patients are randomized to the standard of care arm and participate in all aspects of the study but receive no intervention.
- Physicians (Other): Physicians receive the intervention approximately halfway through data collection for a within subjects, pre-post intervention comparison
  Interventions: Behavioral: Physicians: Educational Module

INTERVENTIONS:
Behavioral: Patients: Questions to Ask Your Doctor: A Workbook for Patient-Doctor Teams — This booklet encourages patients to view themselves as members of the patient-doctor team and to participate actively during clinical interactions by asking questions and stating concerns.
  Arms: Patients--Intervention
Behavioral: Physicians: Educational Module — Physicians will participate in an educational module and receive email prompts to encourage them to discuss trials with all patients who are eligible for a clinical trial, using patient-centered communication
  Arms: Physicians

SUMMARY:
This research has the overall goal of increasing rates at which African American and White men with prostate cancer make an informed decision to participate in a cancer clinical trial.

DETAILED DESCRIPTION:
This research utilizes two distinct research designs to evaluate two separate behavioral interventions.

The first is a between-subject randomized controlled trial to evaluate a patient-focused intervention. The intervention consists of a booklet designed to encourage patients to view themselves as part of the patient-physician team and to participate actively in clinical interactions by asking questions and stating concerns.

The second is a within-subject interrupted time series design to evaluate a physician-focused intervention. The intervention is an educational module and email reminders designed to encourage physicians to discuss trials with all eligible patients using patient-centered communication.In the patient-focused intervention, patients are randomized to an intervention or usual care group, and comparison of outcomes is made between groups.

ELIGIBILITY:
Physician participants

Inclusion criteria:

* Treat patients with prostate cancer
* Able to recruit patients to clinical trials

Exclusion criteria:

* Do not treat patients with prostate cancer
* Not able to recruit patients to clinical trials

Patient Participants

Inclusion criteria:

* Black, African American or White; Non-hispanic confirmed diagnosis of prostate Cancer
* Seeing a participating physician for less than a year and expect to see this physician at least once in the coming year
* Able to read and write English well enough to understand and sign consent forms and respond to questionnaires

Exclusion criteria:

* Not black, African American or White; non Hispanic
* No confirmed diagnosis of prostate cancer
* Not seeing a participating physician or seeing a participating physician for > than one year
* Not able to read and write English well enough to understand and sign consent forms and respond to questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Eggly, Ph.D., Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- [Derived] Eggly S, Manning M, Senft N, Moore TF, Albrecht TL, Penner LA, Heath E, Carducci MA, Lansey DG, Hamel LM. Development and pilot test of a physician-focused cancer clinical trials communication training intervention. PEC Innov. 2021 Dec 16;1:100012. doi: 10.1016/j.pecinn.2021.100012. eCollection 2022 Dec. PMID 37364021
- [Derived] Eggly S, Hamel LM, Heath E, Manning MA, Albrecht TL, Barton E, Wojda M, Foster T, Carducci M, Lansey D, Wang T, Abdallah R, Abrahamian N, Kim S, Senft N, Penner LA. Partnering around cancer clinical trials (PACCT): study protocol for a randomized trial of a patient and physician communication intervention to increase minority accrual to prostate cancer clinical trials. BMC Cancer. 2017 Dec 2;17(1):807. doi: 10.1186/s12885-017-3804-5. PMID 29197371

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 289 patients consented and completed baseline requirement. Of these, 54 qualified for randomization.
Groups:
- Patients Enrolled Not Randomized: Patients enrolled in the trial but did not qualify for randomization
Period: Overall Study
Arm/Group | Patients--Intervention | Patients--Usual Care | Physicians | Patients Enrolled Not Randomized
Started | 25 | 29 | 27 | 235 (Total number of patients 289 minus the number qualified for randomization (54))
Completed | 25 | 29 | 19 | 235
Not Completed | 0 | 0 | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients--Intervention | Patients--Usual Care | Physicians | Total
Number analyzed (Participants) | 25 | 29 | 27 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 25 | 48
  >=65 years | 14 | 17 | 2 | 33
Age, Continuous [Mean (Standard Deviation); unit: years]
  Patients | 66.2 (8.9) | 66.52 (7.6) | 0 (0) | 66.36 (8.15)
  Physicians | 0 (0) | 0 (0) | 47.58 (11.61) | 47.58 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 4
  Male | 25 | 29 | 23 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 13 | 10 | 2 | 25
  White | 12 | 17 | 19 | 48
  Other | 0 | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 27 | 81

OUTCOME MEASURES:

1. Primary Outcome: Physician Offers of a Clinical Trial
Description: Single item: Did the physician offer a trial?
Time Frame: Day of clinical interaction; up to 2 years following enrollment
Population: Data were collected only from participants in the Intervention Group in Phase 1 for this outcome measure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention and Offer: Patients who received the intervention and offer of a trial
Arm/Group | Intervention and Offer
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Patient Decisions to Enroll in a Trial
Description: Single item: Did you agree to participate in this trial?
Time Frame: 1 week following clinical interaction
Reporting Status: Not Posted

3. Secondary Outcome: Patient Active Participation
Description: Observers' global assessment of patients' participation in the interaction
Time Frame: Day of clinical interaction; up to 2 years following enrollment
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Informed Consent (Modified)
Description: 12-item patient-self report on Quality of Informed Consent (QUIC)
Time Frame: 1 week following clinical interaction
Reporting Status: Not Posted

5. Secondary Outcome: Patient Enrollment in Trial
Description: medical chart abstraction
Time Frame: 3 months following clinical interaction
Reporting Status: Not Posted

6. Secondary Outcome: Physician Patient-Centered Communication
Description: Observers' rating of physician communication
Time Frame: Day of clinical interaction; up to 2 years following enrollment
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Trial-Related Communication
Description: Observers' assessment of physician communication related to clinical trials
Time Frame: Day of clinical interaction; up to 2 years following enrollment
Reporting Status: Not Posted

8. Secondary Outcome: Physician Patient-Centeredness
Description: 14-item patient self-report scale
Time Frame: Immediately following clinical interaction
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Patients--Intervention | Patients--Usual Care | Physicians
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02906241/Prot_SAP_000.pdf